CLINICAL TRIAL: NCT05555511
Title: Perioperative Use of N-acetylcysteine to Prevent Acute Kidney Injury in Patients With Pre-existing Moderate Renal Insufficiency Following Cardiac Surgery
Brief Title: Perioperative Use of NAC to Prevent AKI in Patients With Pre-existing Moderate Renal Insufficiency Following Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Alaaeldin Abdelmoneem Alhadidy, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU R 122/2022
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Kidney Injury, Acute
Keywords: N-acetylcysteine; Acute kidney injury; Cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients will be randomized using computer generated random series into two groups according to the used drug into:
  Group A: N-acetylcysteine group (23 Patients) Patients will receive N-acetylcysteine 600 mg intravenous(IV) every 12 hours 24 hours before surgery and will be continued for 48 hours after surgery.
  Group B : Standard (control) group (23 Patients) Patients will not receive N-Acetylcysteine and will receive standard care according to our institutional protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine group (Active Comparator): (23 Patients) Patients will recieve N-acetylcysteine 600 mg intravenous(IV) every 12 hours 24 hours before surgery and will be continued for 48 hours after surgery
  Interventions: Other: Control Group
- Standard group (No Intervention): Patients will not receive N-Acetylcysteine and will receive standard care according to our institutional protocol

INTERVENTIONS:
Other: Control Group — Patients will not receive N-Acetylcystiene and will receive standard care according to our institutional protocol
  Arms: N-acetylcysteine group

SUMMARY:
Acute kidney injury (AKI) or renal impairment is an established complication of cardiac surgery occurring with an incidence up to 30%, To date, no agent has conferred renal protection. Considerable interest has developed in the potential for Nacetylcysteine (NAC) to exert a renoprotective effect in patients undergoing cardiac surgery. Due to the beneficial effect of NAC on contrast nephropathy and its reported anti-inflammatory effects.

DETAILED DESCRIPTION:
Acute kidney injury (AKI), is a well-known complication of cardiac surgery, with an incidence of up to 30% depending on the definition. AKI caused by cardiac surgery is the second most common cause of AKI in the intensive care unit and is a common and serious postoperative complication of cardiac surgery requiring cardiopulmonary bypass (CPB).

The pathogenesis of AKI after CPB is multifactorial, and is mostly due to hypo perfusion, reperfusion injury, activation of the systemic inflammatory response, and/or low cardiac output. Reperfusion will result in the formation of reactive oxygen species, resulting in injury to tissues.

The activation of the systemic inflammatory response is mostly due to the exposure of blood to the extracorporeal CPB circuit, resulting in the activation of the immune system, which is also mediated by the generation of reactive oxygen species. This results in increased recruitment of neutrophils, macrophages, and lymphocytes into the renal parenchyma, leading to AKI.

N-acetylcysteine (NAC) is well known for its antioxidant and free-radical scavenging properties, as well as its vasodilator properties. Its antioxidant properties enable it to prevent ischemic cell death, and as a free-radical scavenger, NAC mitigates the effect of increased reactive oxygen species caused by reperfusion. Hence, theoretically, NAC is able to counteract several mechanisms of kidney injury during cardiac surgery, namely, the systemic inflammatory response, free-radical injury, and ischemia.

In this study, we aimed to investigate if the perioperative use of acetylcysteine will prevent kidney injury after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria

* Scheduled for open heart Surgery with cardiopulmonary bypass (CPB) pump.
* Pre-existing moderate renal insufficiency serum creatinine more than 1.5 mg/dL

Exclusion Criteria:

* Patients on hemodialysis preoperatively
* History of renal transplantation
* IV contrast within 4 days prior to surgery
* Urgent/emergent surgery
* Preoperative hemodynamic instability (intra-aortic balloon pump support or vasoactive medications)
* Planned off-pump surgery;
* Planned deep-hypothermic-circulatory-arrest
* known or suspected allergy to NAC
* Patient Refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-01-26 (Estimated); Study Completion 2023-02-26 (Estimated)

PRIMARY OUTCOMES:
Serum Creatinine rise | 7days
  Creatinine increase >25% or ≥ 0.5 mg/dl above baseline

SECONDARY OUTCOMES:
RRT | 7 days
  Need for Renal Replacement Therapy
Length of ICU stay | 3 days
  Length of stay in the ICU in days
Length of hospital stay | 7 to 10 Days
  Length of stay in hospital in days
Mortality | 30 days
  Mortality rate
Adverse effects | 2 days
  Occurrence of NAC adverse effects as (bronchospasm, urticaria, facial edema, nausea/vomiting).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Alhadidy, Principal Investigator — Ain Shams University
Locations (1):
- Cardiothoracic Academy, Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SH, Kim SJ, Kim HJ, Son JS, Lee R, Yoon TG. Acute Kidney Injury Following Cardiopulmonary Bypass in Children - Risk Factors and Outcomes. Circ J. 2017 Sep 25;81(10):1522-1527. doi: 10.1253/circj.CJ-17-0075. Epub 2017 May 17. PMID 28515370
- [Background] Schopka S, Diez C, Camboni D, Floerchinger B, Schmid C, Hilker M. Impact of cardiopulmonary bypass on acute kidney injury following coronary artery bypass grafting: a matched pair analysis. J Cardiothorac Surg. 2014 Jan 18;9:20. doi: 10.1186/1749-8090-9-20. PMID 24438155
- [Background] Dexter F. Duration of cardiopulmonary bypass and outcome. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):e19; author reply e19-20. doi: 10.1053/j.jvca.2011.12.012. Epub 2012 Jan 29. No abstract available. PMID 22285125
- [Background] Nadim MK, Forni LG, Bihorac A, Hobson C, Koyner JL, Shaw A, Arnaoutakis GJ, Ding X, Engelman DT, Gasparovic H, Gasparovic V, Herzog CA, Kashani K, Katz N, Liu KD, Mehta RL, Ostermann M, Pannu N, Pickkers P, Price S, Ricci Z, Rich JB, Sajja LR, Weaver FA, Zarbock A, Ronco C, Kellum JA. Cardiac and Vascular Surgery-Associated Acute Kidney Injury: The 20th International Consensus Conference of the ADQI (Acute Disease Quality Initiative) Group. J Am Heart Assoc. 2018 Jun 1;7(11):e008834. doi: 10.1161/JAHA.118.008834. No abstract available. PMID 29858368
- [Background] Ates B, Abraham L, Ercal N. Antioxidant and free radical scavenging properties of N-acetylcysteine amide (NACA) and comparison with N-acetylcysteine (NAC). Free Radic Res. 2008 Apr;42(4):372-7. doi: 10.1080/10715760801998638. PMID 18404536
- [Background] Nigwekar SU, Kandula P. N-acetylcysteine in cardiovascular-surgery-associated renal failure: a meta-analysis. Ann Thorac Surg. 2009 Jan;87(1):139-47. doi: 10.1016/j.athoracsur.2008.09.026. PMID 19101287
- [Background] Savluk OF, Guzelmeric F, Yavuz Y, Cevirme D, Gurcu E, Ogus H, Orki T, Kocak T. N-acetylcysteine versus Dopamine to Prevent Acute Kidney Injury after Cardiac Surgery in Patients with Preexisting Moderate Renal Insufficiency. Braz J Cardiovasc Surg. 2017 Jan-Feb;32(1):8-14. doi: 10.21470/1678-9741-2016-0028. PMID 28423123
- [Background] Kotlyar E, Keogh AM, Thavapalachandran S, Allada CS, Sharp J, Dias L, Muller D. Prehydration alone is sufficient to prevent contrast-induced nephropathy after day-only angiography procedures--a randomised controlled trial. Heart Lung Circ. 2005 Dec;14(4):245-51. doi: 10.1016/j.hlc.2005.06.007. Epub 2005 Oct 3. PMID 16360994
- [Background] Diaz-Sandoval LJ, Kosowsky BD, Losordo DW. Acetylcysteine to prevent angiography-related renal tissue injury (the APART trial). Am J Cardiol. 2002 Feb 1;89(3):356-8. doi: 10.1016/s0002-9149(01)02243-3. No abstract available. PMID 11809444